CLINICAL TRIAL: NCT03101644
Title: Optimization of Darunavir Therapy Through Population Pharmacokinetic Modeling, Simulations and Dosage Guidelines
Brief Title: Optimization of Darunavir Therapy and Dosage Recommendations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Laure Elens, Professor, Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UCL-LB-02
Record Dates: First submitted 2017-03-23; First posted 2017-04-05 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Human Immunodeficiency Virus I Infection
MeSH Terms: interventions — Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Darunavir (Other): All patients treated with darunavir
  Interventions: Drug: Darunavir

INTERVENTIONS:
Drug: Darunavir — The investigated drugs are Prezista (darunavir 600 mg twice-daily or 800 mg once-daily) and Rezolsta (darunavir 800 mg/cobicistat 150 mg once-daily)
  Other Names: Prezista; Rezolsta

SUMMARY:
This study will assess and characterize the variability observed in the response to darunavir therapy, an antiretroviral medication used against the Human Immunodeficiency Virus (HIV). More specifically, it aims to quantify variations in the drug's blood concentrations and determine the sources of such variability, both genetic and non-genetic. In light of this information, current dosage guidelines will then be reviewed.

DETAILED DESCRIPTION:
Data will be used to create a population pharmacokinetic model. Inter- and intra-individual pharmacokinetic variability will be quantified and linked to patient-specific covariates, both genetic and non-genetic in nature. Pharmacokinetic-pharmacodynamic relationships will be established, linking drug exposure to efficacy (as measured by CD4 cell count and viral load reduction) and toxicity (as measured by frequency and degree of adverse events). Simulations will be conducted for specific patient profiles and current dosage guidelines reviewed.

Pharmacokinetic design : combined sparse/intensive sampling

* Sparse sampling : One blood sample collected in each individual at a random post-intake time (during a routine visit to the hospital), up to three times over the course of the study period (months 1-18).
* Intensive sampling : Eight blood samples collected over six hours in a subset of twelve individuals (during an additional observation period, months 19-22).

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent
* HIV-positive
* Routinely followed at the Cliniques universitaires Saint-Luc
* Treated with darunavir

Inclusion Criteria (intensive sampling):

- Perfect adherence to treatment (as assessed by anamnesis and based on available PK data for each patient)

Exclusion Criteria:

- N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Darunavir clearance | Up to 18 months (blood sampling for PK once at each visit, three visits per patient over the study period)
  Assessment of darunavir whole-body clearance and inter-compartmental clearance through population pharmacokinetic methods
Darunavir volume of distribution | Up to 18 months (blood sampling for PK once at each visit, three visits per patient over the study period)
  Assessment of darunavir volume of distribution through population pharmacokinetic methods
Darunavir absorption rate | Up to 18 months (blood sampling for PK once at each visit, three visits per patient over the study period)
  Assessment of darunavir absorption rate through population pharmacokinetic methods
Darunavir area under the concentration-time curve (AUC) | Up to 18 months (blood sampling for PK once at each visit, three visits per patient over the study period)
  Assessment of darunavir area under the concentration-time curve through population pharmacokinetic methods
Darunavir maximum plasma concentration (Cmax) | Up to 18 months (blood sampling for PK once at each visit, three visits per patient over the study period)
  Assessment of darunavir maximum plasma concentration through population pharmacokinetic methods

SECONDARY OUTCOMES:
Frequency of adverse events/laboratory abnormalities | Up to 18 months
  Assessment of the frequency of adverse events or laboratory abnormalities
Change in viral load | Up to 18 months
  Assessment of the change in viral load (HIV copies/ml of blood)
Change in blood Cluster of Differentiation 4 (CD4+) T lymphocyte count | Up to 18 months
  Assessment of the change in blood CD4+ T lymphocyte count
Ritonavir/cobicistat AUC | Up to 18 months (blood sampling for PK once at each visit, three visits per patient over the study period)
  Assessment of the pharmacokinetic booster (either ritonavir or cobicistat, depending on the subject) AUC through population pharmacokinetic methods

CONTACTS AND LOCATIONS:
Overall Officials: Leila Belkhir, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stillemans G, Belkhir L, Vandercam B, Vincent A, Haufroid V, Elens L. Exploration of Reduced Doses and Short-Cycle Therapy for Darunavir/Cobicistat in Patients with HIV Using Population Pharmacokinetic Modeling and Simulations. Clin Pharmacokinet. 2021 Feb;60(2):177-189. doi: 10.1007/s40262-020-00920-z. PMID 32696441